CLINICAL TRIAL: NCT00946517
Title: Impaired Family Dynamics Leads to Non Compliance in Type I Diabetes
Status: Terminated | Type: Observational
Why Stopped: PI left the institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB09-00224
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parents: Parents or caregivers of type 1 diabetics
  Interventions: Other: Questionnaires
- Child: Type 1 diabetics
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Parenting and behavioral questionnaires

SUMMARY:
This study will test the hypothesis that certain parenting styles are associated with greater non-adherence to therapy in children and teens with type 1 diabetes. To test their hypothesis, the investigators will use standardized and validated questionnaires for parents and children to determine: parenting styles (the investigators will measure parental strictness, parental attachment, and parental monitoring), parent ability to cope with stress, parent comfort with the parenting role, parent and child level of depression and parent perception of financial resources. The investigators will also measure parent and child's perception of the child's underlying temperament and parent-child conflict. The investigators will correlate these findings with both parent and child subjective measures of adherence to therapy. The investigators will also obtain objective measures of therapy adherence including: HbA1c, number of hospitalizations for diabetes ketoacidosis and number of missed outpatient appointments. These measures will be correlated with our other findings.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetics
* Aged 9 - 18 years

Exclusion Criteria:

* None

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Endocrinology clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Parenting styles | Baseline

SECONDARY OUTCOMES:
Child behavior traits | Baseline
Adherence to therapy | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital, The Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States